CLINICAL TRIAL: NCT02128763
Title: Dry Eye Assessment and Management Study
Acronym: DREAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UPenn IRB Protocol 816490; U10EY022879 (NIH); U10EY022881 (NIH)
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 supplements (Experimental): Total 2000 mg EPA and 1000 mg DHA per day taken in 5 gelcaps
  Interventions: Drug: Omega-3 supplements
- Placebo (Placebo Comparator): Olive oil-5 gelcaps per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3 supplements — 2000 mg EPA and 1000 mg DHA per day
  Arms: Omega-3 supplements
Drug: Placebo — Olive oil gelcaps manufactured to mimic Omega-3 gelcaps
  Arms: Placebo

SUMMARY:
The objective of the DREAM study is to evaluate the effectiveness and safety of supplementation with omega-3 fatty acids in relieving the symptoms of moderate to severe dry eye disease.

DETAILED DESCRIPTION:
The study is designed to:

* Test the hypothesis that omega-3 supplementation is an effective treatment for Dry Eye Disease (DED) in Primary Clinical Trial.
* Better understand DED by describing and evaluating a comprehensive set of features of DED and treatment over 12 months of observation in a well-characterized group of patients.
* Determine the effects of extended use and discontinuation of omega-3 through the Extension trial.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 2 of the following 4 signs in the same eye at screening and baseline visits (Same signs must be present at Screening and Baseline visits): Conjunctival staining present greater than or equal to 1 (out of possible score of 6 per eye), Corneal fluorescein staining present greater than or equal to 4 (out of a possible score of 15 per eye), Tear film break up time (TBUT) less than or equal to 7 seconds, Schirmer's test greater than or equal to 1 to less than or equal to 7 mm in 5 minutes.
* Ocular Surface Disease Index (OSDI) score: 25-80 at screening, 21-80 at baseline.
* Symptoms of DED for greater than or equal to 6 months.
* Use of or desire to use artificial tears at least 2 times per day in preceding 2 weeks.
* Ability to swallow large, soft gelcaps

Exclusion Criteria:

* Allergic to ingredients in supplements or placebo
* Contact lens wear
* Pregnant, nursing, or lactating
* Current ocular infection, inflammation, or acute allergic conjunctivitis
* History of: ocular herpetic keratitis, ocular surgery in past 6 months, LASIK surgery, use of glaucoma medicine or surgery for glaucoma, liver disease, atrial fibrillation, hemophilia or bleeding tendencies
* Currently on anticoagulation therapy
* Eyelid abnormalities or extensive ocular scarring
* Use of EPA/DHA supplements in excess of 1200 mg per dayi
* Current use, insufficient washout period, or intent to change specific treatments for dry eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2014-11; Primary Completion 2017-09-05 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Penny A Asbell, MD, Study Chair — University of Tennessee; Maureen G Maguire, PhD, Principal Investigator — University of Pennsylvania
Locations (27):
- United States (27):
  - Stephen Cohen, OD PC, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Milton M. Hom, OD, FAAO, Azusa, California
  - University of California, Berkeley, Berkeley, California
  - Pendleton Eye Center, Oceanside, California
  - Wolstan and Goldberg Eye Associates, Torrance, California
  - Shettle Eye Research, Largo, Florida
  - Eye Care Centers Management, Inc., Morrow, Georgia
  - University of Illinois Hospital & Health Sciences, Chicago, Illinois
  - Price Vision Group, Indianapolis, Indiana
  - KU Eye Center, Prairie Village, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Clinical Eye Research of Boston, Winchester, Massachusetts
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Minnesota Eye Consultants, P.A., Bloomington, Minnesota
  - Mulqueeny Eye Centers, Creve Coeur, Missouri
  - Tauber Eye Center, Kansas City, Missouri
  - Silverstein Eye Centers, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Universtity of Rochester-Flaum Eye Institute, Rochester, New York
  - Oculus Research at Garner at Eyecarecenter, Raleigh, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Northeast Ohio Eye Surgeons, Kent, Ohio
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania
  - Southern College of Optometry, Memphis, Tennessee
  - The Eye Centers of Racine and Kenosha, Racine, Wisconsin

REFERENCES:
- [Result] Bunya VY, Ying GS, Maguire MG, Kuklinski E, Lin MC, Peskin E, Asbell PA; DREAM Study Research Group. Prevalence of Novel Candidate Sjogren Syndrome Autoantibodies in the Dry Eye Assessment and Management (DREAM) Study. Cornea. 2018 Nov;37(11):1425-1430. doi: 10.1097/ICO.0000000000001714. PMID 30161055
- [Result] Daniel E, Maguire MG, Pistilli M, Bunya VY, Massaro-Giordano GM, Smith E, Kadakia PA, Asbell PA; Dry Eye Assessment and Management (DREAM) Study Research Group. Grading and baseline characteristics of meibomian glands in meibography images and their clinical associations in the Dry Eye Assessment and Management (DREAM) study. Ocul Surf. 2019 Jul;17(3):491-501. doi: 10.1016/j.jtos.2019.04.003. Epub 2019 Apr 22. PMID 31022469
- [Result] Oydanich M, Maguire MG, Pistilli M, Hamrah P, Greiner JV, Lin MC, Asbell PA; Dry Eye Assessment and Management Study Research Group. Effects of Omega-3 Supplementation on Exploratory Outcomes in the Dry Eye Assessment and Management Study. Ophthalmology. 2020 Jan;127(1):136-138. doi: 10.1016/j.ophtha.2019.07.009. Epub 2019 Jul 25. PMID 31445751
- [Result] Roy NS, Wei Y, Yu Y, Ying GS, Kuklinski E, Barry B, Maguire MG, Dana R, Brightwell-Arnold M, Asbell PA; for the Dry Eye Assessment and Management (DREAM) Study Group. Conjunctival HLA-DR Expression and Its Association With Symptoms and Signs in the DREAM Study. Transl Vis Sci Technol. 2019 Aug 21;8(4):31. doi: 10.1167/tvst.8.4.31. eCollection 2019 Jul. PMID 31489258
- [Result] Kuklinski EJ, Hom MM, Ying GS, Lin MC, Chapkin RS, Jones R, Moser A, Kim KY, Maguire MG, Asbell PA; DREAM Study Research Group. Associations Between Systemic Omega-3 Fatty Acid Levels With Moderate-to-Severe Dry Eye Disease Signs and Symptoms at Baseline in the Dry Eye Assessment and Management Study. Eye Contact Lens. 2021 Jan 1;47(1):2-7. doi: 10.1097/ICL.0000000000000687. PMID 32097181
- [Result] Berg EJ, Ying GS, Maguire MG, Sheffield PE, Szczotka-Flynn LB, Asbell PA, Shen JF; DREAM Study Research Group. Climatic and Environmental Correlates of Dry Eye Disease Severity: A Report From the Dry Eye Assessment and Management (DREAM) Study. Transl Vis Sci Technol. 2020 Apr 29;9(5):25. doi: 10.1167/tvst.9.5.25. eCollection 2020 Apr. PMID 32821497
- [Derived] Zhong A, Augello P, Asbell P, Ying GS; DREAM Study Research Group. Intereye Agreement in Dry-Eye Signs in the DREAM Study: Implications for Future Dry-Eye Trials. Cornea. 2025 Feb 1;44(2):149-156. doi: 10.1097/ICO.0000000000003605. Epub 2024 Jul 30. PMID 39079754
- [Derived] Lee DC, Guo M, Yu Y, Bunya VY, Asbell P, Ying GS. Two-Year Progression of Dry Eye Disease in Dry Eye Assessment and Management Study. Cornea. 2024 Oct 1;43(10):1231-1237. doi: 10.1097/ICO.0000000000003503. Epub 2024 Feb 22. PMID 38391283
- [Derived] Hashemi MH, Ambrus JL Jr, Shukla AA, Zhu D, Ying GS, Asbell PA; Dry Eye Assessment and Management (DREAM) Study Research Group. Association of Systemic Markers of Inflammation with Signs and Symptoms of Dry Eye Disease and Sjogren's Syndrome in the Dry Eye Assessment and Management (DREAM(c)) Study. Curr Eye Res. 2024 Jun;49(6):574-581. doi: 10.1080/02713683.2024.2312937. Epub 2024 Feb 12. PMID 38345056
- [Derived] Zhao M, Yu Y, Roy NS, Ying GS, Asbell P, Bunya VY. Sex-related differences and hormonal effects in the Dry Eye Assessment and Management (DREAM) study. Br J Ophthalmol. 2023 Dec 18;108(1):23-29. doi: 10.1136/bjo-2022-322238. PMID 36575626
- [Derived] Sutphin JE, Ying GS, Bunya VY, Yu Y, Lin MC, McWilliams K, Schmucker E, Kuklinski EJ, Asbell PA, Maguire MG; Dry Eye Assessment and Management (DREAM) Study Research Group. Correlation of Measures From the OCULUS Keratograph and Clinical Assessments of Dry Eye Disease in the Dry Eye Assessment and Management Study. Cornea. 2022 Jul 1;41(7):845-851. doi: 10.1097/ICO.0000000000002804. Epub 2021 Jul 21. PMID 34294637
- [Derived] Sayegh RR, Yu Y, Farrar JT, Kuklinski EJ, Shtein RM, Asbell PA, Maguire MG; Dry Eye Assessment and Management (DREAM) Study Research Group. Ocular Discomfort and Quality of Life Among Patients in the Dry Eye Assessment and Management Study. Cornea. 2021 Jul 1;40(7):869-876. doi: 10.1097/ICO.0000000000002580. PMID 33290317
- [Derived] Hussain M, Shtein RM, Pistilli M, Maguire MG, Oydanich M, Asbell PA; DREAM Study Research Group. The Dry Eye Assessment and Management (DREAM) extension study - A randomized clinical trial of withdrawal of supplementation with omega-3 fatty acid in patients with dry eye disease. Ocul Surf. 2020 Jan;18(1):47-55. doi: 10.1016/j.jtos.2019.08.002. Epub 2019 Aug 16. PMID 31425752
- [Derived] Szczotka-Flynn LB, Maguire MG, Ying GS, Lin MC, Bunya VY, Dana R, Asbell PA; Dry Eye Assessment and Management (DREAM) Study Research Group. Impact of Dry Eye on Visual Acuity and Contrast Sensitivity: Dry Eye Assessment and Management Study. Optom Vis Sci. 2019 Jun;96(6):387-396. doi: 10.1097/OPX.0000000000001387. PMID 31116166
- [Derived] Asbell PA, Maguire MG, Peskin E, Bunya VY, Kuklinski EJ; Dry Eye Assessment and Management (DREAM(c)) Study Research Group. Dry Eye Assessment and Management (DREAM(c)) Study: Study design and baseline characteristics. Contemp Clin Trials. 2018 Aug;71:70-79. doi: 10.1016/j.cct.2018.06.002. Epub 2018 Jun 6. PMID 29883769
- [Derived] Dry Eye Assessment and Management Study Research Group; Asbell PA, Maguire MG, Pistilli M, Ying GS, Szczotka-Flynn LB, Hardten DR, Lin MC, Shtein RM. n-3 Fatty Acid Supplementation for the Treatment of Dry Eye Disease. N Engl J Med. 2018 May 3;378(18):1681-1690. doi: 10.1056/NEJMoa1709691. Epub 2018 Apr 13. PMID 29652551

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Olive oil-5 gelcaps per day containing a total of 5 grams of refined olive oil
  Placebo: Olive oil gelcaps manufactured to mimic Omega-3 gelcaps
Period: Overall Study
Arm/Group | Omega-3 Supplements | Placebo
Started | 349 | 186
Completed | 329 | 170
Not Completed | 20 | 16
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 19 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Supplements | Placebo | Total
Number analyzed (Participants) | 349 | 186 | 535
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (13.5) | 57.5 (12.6) | 58.0 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284 | 150 | 434
  Male | 65 | 36 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 24 | 68
  Not Hispanic or Latino | 302 | 161 | 463
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 12 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 25 | 64
  White | 265 | 133 | 398
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 27 | 15 | 42
Region of Enrollment [Number; unit: participants]
  United States | 349 | 186 | 535
OSDI Score [Mean (Standard Deviation); unit: units on a scale] — Ocular Surface Disease Index (OSDI) scores range from 0 to 100, with a score of 0 indicating no ocular discomfort and higher scores indicating greater symptom severity. The minimal clinically meaningful change in score is 10 points.
  units on a scale | 44.6 (14.1) | 44.1 (14.6) | 44.1 (14.2)
Brief Ocular Discomfort Inventory (BODI) Score [Mean (Standard Deviation); unit: units on a scale] — Brief Ocular Discomfort Inventory (BODI) scores range from 0-100. Higher scores = more discomfort. Baseline score is the mean of the screening and eligibility confirmation visit scores.
  units on a scale | 33.2 (15.5) | 33.4 (16.3) | 33.2 (15.8)
EPA level in red cells [Mean (Standard Deviation); unit: percentage of total fatty acids] — Baseline measure of Eicosapentaenoic Acid (EPA) (%) in red blood cells
  percentage of total fatty acids | 0.63 (0.43) | 0.56 (0.35) | 0.60 (0.40)
DHA level in red blood cells at baseline [Mean (Standard Deviation); unit: percentage of total fatty acids] — Baseline measure of Docosahexanoic Acid (DHA) (%) in red blood cells
  percentage of total fatty acids | 3.91 (1.17) | 3.85 (1.11) | 3.9 (1.1)
Oleic Acid (OA) level in red cells [Mean (Standard Deviation); unit: percentage of total fatty acids] — Baseline level of Oleic Acid (OA) in red blood cells (%)
  percentage of total fatty acids | 11.11 (1.24) | 11.10 (1.38) | 11.1 (1.3)
Tear Break Up Time (TBUT) [Mean (Standard Deviation); unit: seconds] — Baseline scores = the average of the screening and baseline visits. Tear Break Up Time (TBUT) is a sign of dry eye disease. Scores range between 0-20 seconds; higher is better.
  seconds | 3.1 (1.4) | 3.1 (1.6) | 3.1 (1.5)
Schimer's Test [Mean (Standard Deviation); unit: mm] — The Schirmer's test determines whether the eye produces enough tears to keep the eye moist. Schirmer's test score range between <4 to >/= to 15 mm of wetting by tears per 5 minutes. Lower scores indicate more severe dry eye.
  mm | 9.3 (6.2) | 10.2 (7.0) | 9.8 (7.2)
Conjunctival Staining [Mean (Standard Deviation); unit: units on a scale] — Instilling a solution into the eye and observing the staining that occurs makes visible any injury or pathology to the ocular surface. Conjunctival staining scores range between 0-6. Lower scores are better (less abnormality).
  units on a scale | 3.1 (1.4) | 2.9 (1.4) | 3.0 (1.4)
Corneal Staining [Mean (Standard Deviation); unit: point score] — Instilling a solution into the eye and observing the staining that occurs makes visible any injury or pathology to the ocular surface. Corneal staining scores range between 0-15. Lower scores are better (less abnormality).
  point score | 4.0 (2.9) | 3.7 (2.4) | 3.9 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Mean of Change From Baseline in Ocular Surface Disease Index (OSDI) Score at 6 and 12 Months
Description: Average of Ocular Surface Disease Index (OSDI) scores from 6 and 12 months minus average of values from screening and eligibility confirmation visits. OSDI scores range from 0 to 100, with a score of 0 indicating no ocular discomfort and higher scores indicating greater symptom severity. The minimal clinically meaningful change in score is 10 points.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo (5 Gms of Refined Olive Oil/Day): Olive oil-5 gelcaps per day
  Placebo: Olive oil gelcaps manufactured to mimic Omega-3 gelcaps
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
units on a scale | -13.9 (15.6) | -12.5 (18.2)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.40, Regression, Linear — P value refers to difference between group on change in overall OSDI score (Row 1)

2. Secondary Outcome: Greater Than or Equal to 10 Point Decrease in Ocular Surface Disease Index (OSDI) (at Least 10 Point Improvement in Symptoms)
Description: Number of participants with at least a 10 point decrease from baseline in Ocular Surface Disease Index (OSDI). Change is the average score at 6 and 12 months minus the average score at the screening and eligibility confirmation visits. OSDI scores range from 0 to 100, with a score of 0 indicating no ocular discomfort and higher scores indicating greater symptom severity. A negative change score = improvement.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (5 Gms of Refined Olive Oil/Day): Olive oil-5 gelcaps per day (5 gms of refined olive oil/day)
  Placebo: Olive oil gelcaps manufactured to mimic Omega-3 gelcaps
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
Participants | 202 | 91
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.09, Regression, Linear

3. Secondary Outcome: Change in Brief Ocular Discomfort Index (BODI) Pain Interference Subscale
Description: Brief Ocular Discomfort Index (BODI) Pain Interference subscale scores range from 0 to 100, with higher scores indicating greater discomfort. Change is the average score at 6 and 12 months minus the average score at the screening and eligibility confirmation visits. A negative change score = improvement.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo (5 Gms Refined Olive Oil/Day): Olive oil-5 gelcaps per day
  Placebo: Olive oil gelcaps manufactured to mimic Omega-3 gelcaps
Arm/Group | Omega-3 Supplements | Placebo (5 Gms Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
score on a scale | -9.4 (15.0) | -8.9 (16.2)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms Refined Olive Oil/Day); Test type: Superiority; p = 0.77, Regression, Linear; Pos hoc application of the Benjamini-Hochberg adjustment

4. Secondary Outcome: Change From Baseline in SF-36 Physical Health Subscale
Description: Medical Outcomes Study 36--Item Short Form Health Survey (SF-36) Physical Health Subscale. Subscale range is 0-100, with higher scores indicating better self reported physical health-related quality of life. Change is the average score at 6 and 12 months minus the average score at the screening and eligibility confirmation visits. A positive change score = improvement.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
score on a scale | 0.1 (6.9) | 0.1 (6.3)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.95, Regression, Linear

5. Secondary Outcome: Change From Baseline in SF-36 Mental Health Subscale
Description: Medical Outcomes Study 26--Item Short Form Health Survey (SF-36) Mental Health Subscale. Mental Health subscale range is 0-100 with higher scores indicating better self reported mental health. Change is the average score at 6 and 12 months minus the average score at the screening and eligibility confirmation visits. A positive change score = improvement.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
score on a scale | -0.9 (6.3) | 0.4 (7.0)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.051, Regression, Linear

6. Secondary Outcome: Compliance With the Study Treatment Protocol as Measured by Change in Blood Levels of EPA
Description: Change in EPA levels in red blood cells - percentage points. Change is the average level at 6 and 12 months minus the level at the eligibility confirmation visit. (Blood was not drawn at the screening visit.) If subjects are compliant, higher EPA levels in red blood cells in the Omega 3 group are expected and no change is expected in the placebo group. Data are missing for 20 subjects in the Omega 3 group and 15 subjects in the placebo group because blood was not drawn at the visit.
Time Frame: 12 months
Population: Data are missing for 20 subjects in the Omega 3 group and 15 subjects in the placebo group.
Measure: Mean (Standard Deviation); unit: percentage of fatty acids in blood cells
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 309 | 155
percentage of fatty acids in blood cells | 2.2 (1.2) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p < 0.001, Regression, Linear

7. Secondary Outcome: Compliance With the Study Treatment Protocol as Measured by Change in Blood Levels of DHA
Description: Change in DHA levels in red blood cells - percentage points. Change is the average score at 6 and 12 months minus the average score at eligibility confirmation visit (blood was not drawn at the screening visit. If compliant, higher DHA levels in red blood cells in the Omega 3 group is expected and no change is expected in the placebo group. Data are missing for 20 subjects in the Omega 3 group and 15 subjects in the placebo group.
Time Frame: 12 months
Population: Data are missing for 20 subjects in the Omega 3 group and 15 subjects in the placebo group.
Measure: Mean (Standard Deviation); unit: percentage of fatty acids in blood cells
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 309 | 155
percentage of fatty acids in blood cells | 1.6 (1.2) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p < 0.001, Regression, Linear

8. Secondary Outcome: Compliance With the Study Treatment Protocol as Measured by Change in Blood Levels of Oleic Acid
Description: Change in Oleic Acid (from olive oil) levels in red blood cells - percentage points. Change is the average score at 6 and 12 months minus the average score at eligibility confirmation visit. (Blood was not drawn at the screening visit.) Data are missing for 20 subjects in the Omega 3 group and 15 subjects in the placebo group because blood was not drawn.
Time Frame: 12 months
Population: Data are missing for 20 subjects in the Omega 3 group and 15 subjects in the placebo group
Measure: Mean (Standard Deviation); unit: percentage of oleic acid in blood cells
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 309 | 155
percentage of oleic acid in blood cells | -0.1 (1.0) | -0.1 (1.0)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.40, Regression, Linear

9. Secondary Outcome: Change in Conjunctival Staining Score
Description: Average change from 6 and 12 months minus average of values from screening and eligibility confirmation visits among eyes that qualified for the study. Scores range between 0-6, with higher scores indicate more severity. A negative change indicates improvement.
Time Frame: 12 months
Population: Among eyes that qualified for the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
Number analyzed (eyes) | 629 | 327
units on a scale | -0.4 (1.1) | -0.4 (1.0)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.77, Regression, Linear

10. Secondary Outcome: Change in Schirmer's Test mm
Description: The Schirmer's test measures the production of tears by an eye as measured by mm of wetting of a strip of paper attached to the lower lid for 5 minutes. Scores range from 0 to 30 or more mm. Lower scores indicate more severe dry eye. Change is the average change from 6 and 12 months minus average of values from screening and eligibility confirmation visits among eyes that qualified for the study.
Time Frame: 12 months
Population: among eligible eyes
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
Number analyzed (eyes) | 629 | 327
mm | 0.4 (5.3) | 0.3 (5.0)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.95, Regression, Linear

11. Secondary Outcome: Change in Tear Film Break up Time, in Seconds
Description: Average of values from 6 and 12 months minus average of values from screening and eligibility confirmation visits. Possible range of scores is 0->20. Low values indicate greater severity. A positive change score = improvement.
Time Frame: 12 months
Population: Measure is eyes, not people.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
Number analyzed (eyes) | 629 | 327
seconds | 0.7 (2.1) | 0.6 (1.6)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.25, Regression, Linear

12. Secondary Outcome: Change in Corneal Fluorescein Staining Score
Description: Average change from 6 and 12 months minus average of values from screening and eligibility confirmation visits among eyes that quality that qualified for the study. Possible range of scores is 0-15; higher scores indicate more severity. A negative change indicates improvement.
Time Frame: 12 months
Population: Average change from 6 and 12 months minus average of values from screening and eligibility confirmation visits among eyes that quality that qualified for the study
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
Number analyzed (eyes) | 629 | 327
units on a scale | -0.6 (1.9) | -0.7 (1.7)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.61, Regression, Linear

13. Secondary Outcome: Change in Visual Acuity
Description: Visual acuity scores of 0-100 correspond to Snellen visual acuity levels of worse than 20/800 to 20/10, respectively. Higher change score = improved visual acuity.
Time Frame: 12 months
Population: Each eye measured separately. Total are numbers of eyes assessed, not subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 329 | 170
Number analyzed (eyes) | 656 | 340
score on a scale | -0.5 (5.0) | -0.2 (4.8)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.42, Regression, Linear

14. Secondary Outcome: Change in Use of Artificial Tears and Other Treatments for Dry Eye Disease
Description: Subjects with change in number of treatments used for dry eye disease, n.,(%)
Time Frame: 12 months
Population: Data are missing for 5 subjects in the omega -3 group and 6 subjects in the placebo group
Measure: Count of Participants; unit: Participants
Arm/Group | Omega-3 Supplements | Placebo (5 Gms of Refined Olive Oil/Day)
Number analyzed (Participants) | 324 | 164
Participants
  Fewer treatments used, with no additions | 171 | 93
  No Change | 80 | 36
  ≤ treatments used, with ≥1 treatment switched | 40 | 23
  More treatments used | 33 | 12
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms of Refined Olive Oil/Day); Test type: Superiority; p = 0.60, Chi-squared, Corrected

15. Other Pre Specified Outcome: Change in Intraocular Pressure (IOP)- mm Hg
Description: Eye pressure is measured in millimeters of mercury (mm Hg). Normal eye pressure ranges from 12-22 mm Hg, and eye pressure of greater than 22 mm Hg is considered higher than normal. Included as a safety measure.
Time Frame: 12 months
Population: Each eye measured separately
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo
Number analyzed (Participants) | 329 | 170
Number analyzed (eyes) | 658 | 340
mmHg | 0.0 (2.3) | 0.3 (2.4)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo; Test type: Superiority; p = 0.17, Regression, Linear

16. Other Pre Specified Outcome: Change in Tear Break up Time by Keratography
Description: Tear breakup time (TBUT) is used to assess for evaporative dry eye disease. In this measure, TBUT is measured using the keratograph machine. TBUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film. Change is the average of values from 6 and 12 months minus average of values from screening and eligibility confirmation visits.
Time Frame: 12 months
Population: Each eye is measured separately. Total are number of eyes assessed, not subjects. Tear Break up Time by Keratography was only measured at the 13 clinical centers that owned an Oculus Keratograph machine; therefore the number of participants analyzed for this measure is less than the overall number of study participants.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo (5 Gms Refined Olive Oil/Day)
Number analyzed (Participants) | 154 | 80
Number analyzed (eyes) | 290 | 149
seconds | -0.5 (6.7) | -0.5 (6.1)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms Refined Olive Oil/Day); Test type: Superiority; p = 0.02, Regression, Linear

17. Other Pre Specified Outcome: Change in Tear Meniscus Height( TMH) by Keratography
Description: The purpose of the tear film is to reduce evaporation of natural tears. Assessment of the tear film meniscus is a quantitative measurement of tear film quantity. In this measure, TMH is measured using the keratograph machine. Change is the average of values from 6 and 12 months minus average of values from screening and eligibility confirmation visits.
Time Frame: 12 months
Population: Each eye measured separately. Total are number of eyes assessed, not subjects. Tear Meniscus Height by Keratography was only measured at the 13 clinical centers that owned an Oculus Keratograph machine; therefore, the number of participants analyzed for this measure is less than the overall number of study participants.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo (5 Gms Refined Olive Oil/Day)
Number analyzed (Participants) | 167 | 87
Number analyzed (eyes) | 317 | 162
mm | 0.00 (0.16) | -0.01 (0.14)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms Refined Olive Oil/Day); Test type: Superiority; p = 0.71, Regression, Linear

18. Other Pre Specified Outcome: Change in Redness by Keratography
Description: Change in ocular redness as measured using the keratograph machine. Change is the average of values from 6 and 12 months minus average of values from screening and eligibility confirmation visits. Title of the Scale used to measure outcome: Oculus Keratograph 5M R-scan, Scale Ranges: 0.0-4.0. A lower number indicates a better outcome (less redness).
Time Frame: 12 months
Population: Each eye measured separately. Total are number of eyes assessed, not subjects. Change in redness measured by keratography was only performed at the 13 clinical centers that owned an Oculus Keratograph machine; therefore, the number of participants analyzed for this measure is less than the overall number of study participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo (5 Gms Refined Olive Oil/Day)
Number analyzed (Participants) | 150 | 80
Number analyzed (eyes) | 273 | 145
score on a scale | -0.00 (0.34) | -0.01 (0.40)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms Refined Olive Oil/Day); Test type: Superiority; p = 0.66, Regression, Linear

19. Other Pre Specified Outcome: Change in Tear Osmolarity
Description: Tear osmolarity measures the salt content of the tears. Higher the osmolarity indicate more severe dry eye. Change is the average of values from 6 and 12 months minus average of values from screening and eligibility confirmation visits. A lower change score indicates improvement.
Time Frame: 12 months
Population: Each eye is measured separately. Total are number of eyes assessed, not subjects.Tear Osmolarity was only performed at the 18 clinical centers that owned a Tearlab osmolarity machine; therefore the number of participants analyzed for this measure is less than the overall number of study participants.
Measure: Mean (Standard Deviation); unit: mOsms/L
Units Other Than Participants: eyes
Arm/Group | Omega-3 Supplements | Placebo (5 Gms Refined Olive Oil/Day)
Number analyzed (Participants) | 233 | 117
Number analyzed (eyes) | 424 | 212
mOsms/L | -0.7 (21.5) | 3.6 (18.3)
Statistical Analysis 1: Comparison: Omega-3 Supplements vs Placebo (5 Gms Refined Olive Oil/Day); Test type: Superiority; p = 0.02, Regression, Linear

ADVERSE EVENTS:
Time Frame: AE data were collected from the safety visit to 12 months The AE reporting period was the from the screening visit to the end of the study follow-up (12 months). At the last visit, subjects were instructed to report any subsequent event(s) occurring within 30 days that the subject or a physician, believed might reasonably be related to study treatment. Subjects who withdrew early were contacted by the Clinic Coordinator 30 days after their last visit to ascertain whether any AEs occurred.
Arm/Group | Omega-3 Supplements | Placebo
All-Cause Mortality (participants affected / at risk) | 1/349 | 0/186
Serious Adverse Events (participants affected / at risk) | 21/349 | 15/186
Other Adverse Events (participants affected / at risk) | 0/349 | 0/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Supplements (N=349) | Placebo (N=186)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GALLBLADER PAIN (Hepatobiliary disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
FACIAL PALSY (Nervous system disorders) | 0 (0) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (2) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ARTHRODESIS (Surgical and medical procedures) | 0 (0) | 1 (1)
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 (0) | 2 (2)
COLECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
GASTROINTESTINAL ENDOSCOPIC THERAPY (Surgical and medical procedures) | 1 (1) | 0 (0)
HYSTERECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 1 (1)
OVARIAN CYSTECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
PARATHYROIDECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02128763/Prot_SAP_ICF_000.pdf